CLINICAL TRIAL: NCT02607969
Title: Comparison the Effectiveness Control Frequency of Physiotherapy Home Program on Deformational Plagiocephaly
Brief Title: Investigating the Effectiveness of Control Frequency on and Deformational Plagiocephaly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G014/15
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Deformational Plagiocephaly
Keywords: Deformational Plagiocephaly,Treatment,Compliance
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- seen once every six weeks (Experimental): Parents will be educated about home program and they will be asked to control once every six weeks.
  Interventions: Other: Home program
- seen once a week. (Experimental): Parents will be educated about home program and they will be asked to control once a week.
  Interventions: Other: Home program

INTERVENTIONS:
Other: Home program — Parents will be educated about the home program which consisted of positioning the neck and head, sleep in alternating head positions and in side-laying to increase head shape symmetry and place infants, when awake and under supervision, regularly in the prone position a day to stimulate normal motor development (tummy time), decreasing the time spent in car seat at supine position. Environmental settings also were given to challenge the baby look through from the side no flattening to room, place colorful and sonorous toys or mirror on the opposite of the flattening side, and stimulate active rotation by communicating with baby from this side. Handling strategies, stretching and strengthening exercises will given for CMT

SUMMARY:
30 babies with Deformational Plagiocephaly (DP) due to the congenital muscular torticollis will be the participants of the study.

The subjects will randomly allocated into the two home program groups; first home program group was seen once every six weeks (SxW), second home program group was seen once a week (OW).

Parents will educate about the same home program which consisted of positioning the neck and head, sleep in alternating head positions and in side-laying to increase head shape symmetry and place infants, when awake and under supervision, regularly in the prone position a day to stimulate normal motor development (tummy time), decreasing the time spent in car seat at supine position. Environmental settings also will be given to challenge the baby look through from the side no flattening to room, place colorful and sonorous toys or mirror on the opposite of the flattening side, and stimulate active rotation by communicating with baby from this side. Handling strategies, stretching and strengthening exercises will be given for CMT. The parents will be reinforme if necessary. Positioning strategies will spread throughout the day.Plagiocephaly severity assessment scale (PSS) which has 5 subgroups as following frontal asymmetry, occipital flattening, head tilt, fascial asymmetry, ear asymmetry will be used to evaluate severity of DP.

DETAILED DESCRIPTION:
30 babies with Deformational Plagiocephaly due to the congenital muscular torticollis will be the participants of the study.

The subjects will randomly allocate into the two home program groups; first home program group was seen once every six weeks (SxW), second home program group was seen once a week (OW), by utilizing sealed envelope if babies met the following inclusion and exclusion criteria.

After the initial evaluation, parents will be educate about the same home program which consisted of positioning the neck and head, sleep in alternating head positions and in side-laying to increase head shape symmetry and place infants, when awake and under supervision, regularly in the prone position a day to stimulate normal motor development (tummy time), decreasing the time spent in car seat at supine position. Environmental settings also will be given to challenge the baby look through from the side no flattening to room, place colorful and sonorous toys or mirror on the opposite of the flattening side, and stimulate active rotation by communicating with baby from this side. Handling strategies, stretching and strengthening exercises will be given CMT. One or two days after the first visit the parents will asked to come again and demonstrate how they had implemented the home program and what adaptations they had made. The parents will be reinformed if necessary. Positioning strategies will spread throughout the day.

Participants will be allocated to the groups with sealed envelope randomization after parent will be given the same home program.

ELIGIBILITY:
Inclusion Criteria:

* Babies with congenital muscular torticollis and secondary deformational plagiocephaly
* Head tilt from 5 to 20 degrees
* Age between 0-6 months

Exclusion Criteria:

* Have another health problem such as neurological, vertebral anomalies, craniosynostosis

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
plagiocephaly severity scale | Change from Baseline in head tilt at 6th weeks of treatment, at the end of the treatment/12th weeks, at follow up/18th weeks
  scale which has 5 subgroups as following frontal asymmetry, occipital flattening, head tilt, fascial asymmetry, ear asymmetry.

SECONDARY OUTCOMES:
Head tilt with photographic method | Change from Baseline in head tilt at 6th weeks of treatment, at the end of the treatment/12th weeks, at follow up/18th weeks
  Baby lies supine while taking photo of baby's habitual head position. The angle between the two lines, connecting eyes pupils and connecting acromions, is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal KEKLİCEK, PhD, PT, Principal Investigator — Hacettepe University,Faculty of Health Sciences Department of Physiotherapy